CLINICAL TRIAL: NCT03967249
Title: An Open-Label Extension Trial of IONIS GHR-LRx, an Antisense Inhibitor of the Growth Hormone Receptor Administered Monthly Subcutaneously to Patients With Acromegaly Being Treated With Long-Acting Somatostatin Receptor Ligands (SRL)
Brief Title: Extension Study of IONIS-GHR-LRx Administered to Participants With Acromegaly Being Treated With Long-acting Somatostatin Receptor Ligands
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 766720-CS3; 2019-000591-42 (EudraCT Number)
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Acromegaly
Keywords: Acromegaly, IONIS-GHR-LRx
MeSH Terms: conditions — Acromegaly | interventions — lanreotide; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IONIS GHR-LRx + Somatostatin Receptor Ligand (SRL) (Experimental): IONIS GHR-LRx (as per dose in previous study) will be administered subcutaneously once every 28 days for 53 weeks.
  Interventions: Drug: IONIS GHR-LRx; Drug: Somatostatin Receptor Ligand (SRL)

INTERVENTIONS:
Drug: IONIS GHR-LRx — Participants will receive IONIS GHR-LRx by subcutaneous injection.
Drug: Somatostatin Receptor Ligand (SRL) — Participants will receive Somatostatin Receptor Ligand (lanreotide, octreotide) once monthly.
  Other Names: lanreotide; octreotide

SUMMARY:
The purpose of this study is to assess the safety and efficacy of extended dosing with IONIS GHR-LRx in participants with acromegaly as add-on to somatostatin receptor ligands (SRL) therapy.

DETAILED DESCRIPTION:
This extension study will include participants up to 60 participants with acromegaly from Study NCT03548415. All participants will remain on the same dose from the previous study and receive IONIS GHR-LRx (SC) injection once every 28 days as add-on to SRL therapy for 53 weeks. At the end of 53 weeks, participants will enter a 14-week post-treatment (PT) evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Randomized in index trial (CS2) and completed the entire study, or completion of the treatment period for CS2 and completed or plan to complete PTWK5 visit with an acceptable safety profile, per investigator judgment
* Participants with confirmed stable monthly regimen of SRL for 3 months prior to screening
* Able and willing to participate in a 53-week treatment and 14-week post-treatment study

Exclusion Criteria:

* Treatment with any other acromegaly medications taken prior to Day 1 within the time period: bromocriptine: 2 weeks, carbergoline: 4 weeks, quinagolide: 4 weeks, pegvisomant: 4 weeks and pasireotide: 4 months
* Participant who received surgery for pituitary adenoma in the last 3 months prior to screening and participants needing and/or planning to receive surgery for the pituitary adenoma during the trial
* Unwilling to comply with required study procedures during the treatment and post-treatment periods

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
The Incidence of Adverse Events | Up to approximately 16 months
  Incidence of adverse events (AEs), serious AEs, treatment related AEs, AEs leading to withdrawal

SECONDARY OUTCOMES:
Percent Change from Baselines in Insulin-like Growth Factor I (IGF-1) Levels | Baseline and at Week 26 and Week 53
Percentage of Participants who Achieve Normalized IGF-1 Levels to Within 1.2 Times of Gender and Age-Adjusted Upper Limits | Week 26 and at 28 days after the Week 53 dose
Percentage of Participants who Achieve Normalized IGF-1 Levels to Within 1.0 Times of Gender and Age-Adjusted Upper Limits | Week 26 and at 28 days after the Week 53 dose
Percentage of Participants who Begin Other Acromegaly Medication | Up to approximately 16 months
Time From First Dose of IONIS GHR-LRx in this open label extension (CS3) to Date of Initiation of Other Acromegaly Medications | Up to approximately 16 months

CONTACTS AND LOCATIONS:
Locations (22):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern University, Evanston, Illinois
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
- Magyar Honvedseg Allami Egeszsegugyi Kozpont, II. sz Belgyogyaszat Osztaly, Budapest, Hungary
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences (LSMU) Kauno klinikos - Endocrinology clinic, Kaunas
  - Vaidoto Urbanaviciaus Individuali imone - Endokrinologijos klinika, Vilnius
- Poland (3):
  - Centrum Nowoczesnych Terapii "Dobry Lekarz" Sp. z o. o., Krakow
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Mazowiecki Szpital Brodnowski, Warsaw
- Russia (9):
  - Multi-field Medical Clinic Anturium LLC, Barnaul
  - Interregional Clinical Diagnostic Center, Kazan'
  - Kemerovo Regional Clinical Hospital n.a. S.V. Belyaev, Kemerovo
  - Federal State Budget Institution "National Medical Research Center of Endocrinology" of the Ministry of Healthcare of the Russian Federation, Moscow
  - I.M. Sechenov Moscow First State Medical University, Moscow
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Orenburg Regional Clinical Hospital, Orenburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - State Budget Healthcare Institution of the Tver Region (Regional Clinical Hospital), Tver'
- Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No